CLINICAL TRIAL: NCT03898778
Title: Effects of the Minnesota Medical Technologies Anal Insert Device in Fecal Incontinence
Brief Title: Effects of an Anal Insert Device in Fecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnesota Medical Technologies (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-004642; NCT03934463 (obsolete NCT alias)
Record Dates: First submitted 2019-03-30; First posted 2019-04-02 (Actual); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Fecal Incontinence
Keywords: bowel incontinence; accidental bowel leakage; rectal diseases; intestinal diseases; gastrointestinal diseases; digestive system diseases; diarrhea; loose stool; stool leakage; watery stool; involuntary bowel leakage
MeSH Terms: conditions — Fecal Incontinence; Rectal Diseases; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Subjects with fecal incontinence (Experimental): Male and female subjects aged 18 years and older with a diagnosis of fecal incontinence who have failed conservative medical therapy (i.e., the use of bulking agents, anti-diarrheal agents (e.g., loperamide and biofeedback therapy as appropriate) for fecal incontinence will be treated with an anal insert device.
  Interventions: Device: Minnesota Medical Technologies Anal Insert Device

INTERVENTIONS:
Device: Minnesota Medical Technologies Anal Insert Device — Non-sterile soft, flexible, liquid-filled anal insert either 10 mm size or 13 mm size, meant for single use only

SUMMARY:
The purpose of this research is to test the effects of an inserted anal device on fecal incontinence (accidental bowel leakage) in patients who have persistent symptoms despite other conservative therapy.

DETAILED DESCRIPTION:
This is a prospective, open label study designed to evaluate the efficacy, safety, and tolerability of the Minnesota Medical Technologies Anal Insert Device in participants with Fecal Incontinence (FI).

ELIGIBILITY:
Inclusion Criteria

* Able to provide signed (written) informed consent
* Diagnosis of fecal incontinence, with duration of symptoms six months or longer with a history of at least one fecal incontinence (FI) episode per week or at least four episodes per month
* Subject comprehends study meaning and is capable of carrying out study duties
* Patient is fluent in English as study questionnaires have been validated using English
* If female and of childbearing potential, patient has had a negative urine pregnancy test within 21 days of the first day of the baseline visit
* If applicable, patient agrees to use acceptable birth control (surgical sterilization, abstinence, approved hormonal contraceptives such as birth control pills, barrier methods such as condom or diaphragm used with a spermicide, or an intrauterine device (IUD)). If not applicable, the reason why shall be documented on the screening log.
* Subject is at least 18 years of age at time of consent
* Patients has failed conservative medical therapy (i.e., the use of bulking agents, anti-diarrheal agents (e.g., loperamide) and biofeedback therapy as appropriate) for Fecal Incontinence

Exclusion Criteria

* Unable or unwilling to provide informed consent or to comply with study procedures
* History of anorectal pathology in the past 6 months (perianal abscess or fistula, fecal impaction, or clinically significant rectocele).
* History of inflammatory bowel disease with active proctosigmoiditis
* History of rectal surgery in past 6 months where the Investigator determines that the use of the study device may be associated with an increased risk of complications.
* History of acute or chronic illness or history of illness or any other reason which in the opinion of the Investigator, could pose a threat or harm to the subject or obscure interpretation of laboratory test results or interpretation of study data such as frequent angina, Class III or IV congestive heart failure, etc. The reason for exclusion of any enrolled subject shall be documented on the screening log.
* Patient has known clinically-significant immune deficiency state (e.g., HIV infection).
* Patient is taking drugs with a low therapeutic index, such as warfarin, digoxin, and anti-seizure medications
* If patient has clinically suspected upper or lower gastrointestinal (GI) obstruction, they must be excluded or have been evaluated per standard of care and obstruction ruled out before screening. Determination of obstruction shall be documented on the screening log.
* History of fecal impaction with overflow diarrhea in the past 6 months
* History of Ileo-anal pouch
* History of allergy to silicone or one of its components
* Patient is pregnant and/or nursing
* Any other reason, which in the opinion of the Investigator, would confound proper interpretation of the study
* Patient whom, after training from a healthcare provider, cannot insert or expel the device themself or with assistance from a caregiver
* History of anal or rectal pain and/or rectal bleeding in the past month
* Subject cannot retain either device (10 or 13 mm) while ambulating at the screening visit
* Post baseline anoscopy examination, presence of an anal fissure, Grade III-IV internal hemorrhoids, or thrombosed external hemorrhoids.

In addition, subjects will not be eligible to participate in the Treatment Period if during the baseline period or at the anorectal manometry visit:

* Used rescue medications beyond those allowed by the protocol
* demonstrated lack of compliance (for e.g., did not complete bowel diaries for 3 days in any week during the baseline diary period).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil E Bharucha, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the study was initiated in May 2019 and completed in October 2023. Potential subjects were approached by advertising, letter, phone, in person, or by e-mail.
Period: Overall Study
Arm/Group | Subjects With Fecal Incontinence
Started | 124
Completed | 59
Not Completed | 65

BASELINE CHARACTERISTICS:
Population: ITT population
Arm/Group | Subjects With Fecal Incontinence
Number analyzed (Participants) | 59
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 57
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Primary Effectiveness Endpoint
Description: Percent treatment responders (proportion of subjects with percent relative change of Accidental Bowel Leakage (ABL) ≥ 50%) for the modified Intent to Treat (mITT) population.
Time Frame: Baseline (Weeks 1-4) through Treatment period (Weeks 9-12)
Population: modified Intent to Treat (mITT)
Measure: Number (95% Confidence Interval); unit: percentage of treatment responders
Arm/Group | Subjects With Fecal Incontinence
Number analyzed (Participants) | 58
percentage of treatment responders | 75.9 [62.83 to 86.13]

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 16 weeks.
Arm/Group | Subjects With Fecal Incontinence
All-Cause Mortality (participants affected / at risk) | 0/124
Serious Adverse Events (participants affected / at risk) | 1/124
Other Adverse Events (participants affected / at risk) | 12/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Fecal Incontinence (N=124)
Diastolic dysfunction and relative chronotropic insufficiency (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Fecal Incontinence (N=124)
Leg pain (Injury, poisoning and procedural complications) | 1 (1) — Leg pain from injury slipping in shower diagnosed with thigh contusion
Cough and nasal congestion (Infections and infestations) | 1 (1) — Bronchitis
Anorectal irritation, pain, soreness (Gastrointestinal disorders) | 1 (1) — Preexisting anal fissure identified at time of device fit test prior to fitting period.
Perianal irritation and anorectal discomfort (worsening) (Gastrointestinal disorders) | 1 (1) — Hemorrhoids
Nausea and vomiting (Gastrointestinal disorders) | 1 (1)
Perianal pruritus and soreness (Gastrointestinal disorders) | 1 (1)
Device over-insertion or device migration into anal canal or rectum (Gastrointestinal disorders) | 1 (1)
chest and extremity pain (Injury, poisoning and procedural complications) | 1 (1) — Abrasions, bruising, and fraction of the sternum due to falling off of a ladder.
Dysuria (Gastrointestinal disorders) | 1 (1) — Urinary tract infection
Abdominal cramping (Gastrointestinal disorders) | 1 (1)
Perianal pain and bleeding related to flair of lichen sclerosis (Gastrointestinal disorders) | 1 (1)
Herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Diarrhea and vomiting (Gastrointestinal disorders) | 1 (1) — Gastroenteritis
Abnormal liver function tests (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT03898778/Prot_SAP_001.pdf